CLINICAL TRIAL: NCT07185308
Title: Postbiotics Ameliorate Cancer Cachexia in Patients With Non-small-cell Lung Cancer: a Multicentre, Double-blind, Randomised Controlled Trial
Brief Title: Postbiotics Ameliorate Cachexia in Patients With Non-small-cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); The First Hospital of Jilin University (Other); Fujian Cancer Hospital (Other Government); Zhongnan Hospital (Other); National Cancer Center/National Cancer Clinical Medical Research Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Unknown); Affiliated Hospital of Jiangnan University (Other); Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Henan University (Unknown); Shanghai Changzheng Hospital (Other); Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hongxia Xu, Director of the Department of Clinical Nutrition, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP-2025-239
Record Dates: First submitted 2025-09-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cachexia; Cancer
Keywords: Non-small-cell lung cancer; Cachexixa; Postbiotics
MeSH Terms: conditions — Cachexia; Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo + standard chemotherapy + ICIs (PD-1/PD-L1 inhibitors. The placebo was administered at the same dose and on the same schedule as the JK-5G group.
  Interventions: Dietary Supplement: Placebo, 2.5 g per dose, three times per day
- JK-5G postbiotics group (Experimental): JK-5G + standard chemotherapy + ICIs (PD-1/PD-L1 inhibitors). The intervention period for JK-5G spanned 90 days, covering four 21-day chemotherapy cycles, with a dosage of 2.5 g administered three times daily.
  Interventions: Dietary Supplement: Postbiotics, 2.5 g per dose, three times per day

INTERVENTIONS:
Dietary Supplement: Postbiotics, 2.5 g per dose, three times per day — Postbiotics oral powder, 2.5 g per dose, administered three times daily for a total duration of 90 days (four 21-day chemotherapy cycles).
  Arms: JK-5G postbiotics group
Dietary Supplement: Placebo, 2.5 g per dose, three times per day — Placebo made of cyclodextrine, oral powder, 2.5 g per dose, administered three times daily for a total duration of 90 days (four 21-day chemotherapy cycles).
  Arms: Control group

SUMMARY:
This study aims to evaluate the efficacy of the oral postbiotic preparation JK-5G in improving body weight among patients with non-small-cell lung cancer (NSCLC)-related cachexia. By means of a randomized controlled trial, we will compare the between-group difference in body-weight changes between the JK-5G and placebo arms to clarify its nutritional therapeutic benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender.

   -
2. Patients with histologically or cytologically confirmed non-small-cell lung cancer (NSCLC) classified as stage III-IV according to the 9th TNM edition of IASLC, who are either currently receiving or have completed chemotherapy combined with immunotherapy.

   -
3. Cachexia was diagnosed according to the international consensus criteria: involuntary weight loss >5 % within 6 months preceding screening, or BMI <20 kg/m² combined with >2 % involuntary weight loss within the same period.

   -
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3 and an estimated life expectancy of ≥ 4 months.

   -
5. Prior to the first dose of study treatment, adequate organ function must be documented (no blood products, granulocyte-colony-stimulating factors, or thrombopoietic agents within 14 days before randomisation): 1) Absolute neutrophil count ≥ 1.5 × 10^9/L;2)Platelet count ≥ 100 × 10^9/L; 3) Haemoglobin > 90 g/L; 4) Serum creatinine < 1.5 × upper limit of normal (ULN) or creatinine clearance (Cockcroft-Gault) > 50 mL/min; 5) Total bilirubin < 1.5 × ULN (< 3 × ULN in Gilbert's syndrome) ;6) AST and ALT < 2.5 × ULN (≤ 5 × ULN if hepatic metastases present); 7) INR and aPTT ≤ 1.5 × ULN unless the participant is on therapeutic anticoagulation; 8) Left-ventricular ejection fraction (LVEF) > 50 %

   -
6. Participants must be capable of providing written informed consent and comprehending the potential risks associated with the intervention.

   -
7. Participants must demonstrate high adherence to the study protocol.

   -
8. Gastrointestinal function score of < 5.

Exclusion Criteria:

1. Current presence of reversible causes of reduced food intake (e.g., oral mucositis or mechanical obstruction).

   -
2. Participants who are receiving tube feeding or parenteral nutrition at the time of screening or randomization.

   -
3. Cachexia attributable to other etiologies (e.g., chronic obstructive pulmonary disease, heart failure, or HIV/AIDS).

   -
4. Major surgery within 4 weeks prior to randomization or major surgery planned during the study period.

   -
5. Initiation of systemic corticosteroid therapy within 4 weeks prior to randomization.

   -
6. Use of any appetite- or weight-enhancing agent within 30 days before randomisation, including anamorelin, megestrol acetate, cannabinoids, olanzapine, or mirtazapine.

   -
7. Use of antibiotics or probiotic-containing medications/foods within 2 weeks prior to randomization.

   -
8. Use of glucagon-like peptide-1 (GLP-1) receptor agonists for weight reduction within 30 days prior to randomization.

   -
9. Pregnant or lactating women.

   -
10. Participants who are unable to understand the study objectives or who do not agree to comply with the study requirements.

    -
11. Individuals who lack full legal capacity or whose legal capacity is restricted.

    -
12. Any medical condition that could interfere with the interpretation of study results or increase the participant's risk in the opinion of the investigators.

    -
13. Participation in any other clinical trial.

    -
14. Gastrointestinal function score of ≥ 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Body-weight change | From enrollment to the end of treatment at 12 weeks
  The primary endpoint of this study is the between-group difference in change from baseline to week 12 in body weight between the postbiotics arm and the placebo arm.

SECONDARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 12 weeks
  The week-12 objective response rate evaluated by CT imaging based on RECIST 1.1 criteria
FAACT-ACS score | From enrollment to the end of treatment at 12 weeks
  Change from baseline to week 12 in the FAACT subscale scores (FAACT-ACS and FAACT-5IASS).
MDASI score | From enrollment to the end of treatment at 12 weeks
  Changes from baseline to week 12 in the pain, fatigue, nausea, and sleep disturbance items of the M.D. Anderson Symptom Inventory (MDASI)
Immuno-inflammatory biomarker changes | From enrollment to the end of treatment at 12 weeks
  Biomarker changes in CRP、IL-1、IL-6 and TNF-α
The EORTC Quality-of-Life Questionnaire Core | From enrollment to the end of treatment at 12 weeks
  Changes in the EORTC Quality-of-Life Questionnaire Cores scores, a 30-item cancer-specific instrument that yields five functional scales.
Circulating growth-differentiation factor-15 (GDF-15) levels | From enrollment to the end of treatment at 12 weeks
  Changes in circulating growth-differentiation factor-15 (GDF-15) levels
Incidence of adverse events | From enrollment to the end of treatment at 12 weeks
  Incidence of adverse events and occurrence of laboratory abnormalities, vital-sign anomalies, and electrocardiographic deviations.
Lumbar skeletal muscle index (LSMI) assessed by computed tomography | From enrollment to the end of treatment at 12 weeks
  Change from baseline in lumbar skeletal muscle index (LSMI) assessed by computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Xu, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study results will be made publicly available in the form of academic publications.